CLINICAL TRIAL: NCT00239499
Title: A Six-Week, Randomised, Double-Blind, Triple-Dummy, Parallel Group, Multiple Dose, Pilot Study Comparing Tiotropium Inhalation Capsules to Salmeterol Inhalation Aerosol Combined With Fluticasone Inhalation Aerosol in Patients With Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Pilot Study Comparing Tiotropium (Spiriva) to Salmeterol (Serevent) Plus Fluticasone (Flixotide) in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.273
Record Dates: First submitted 2005-10-14; First posted 2005-10-17 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Salmeterol Xinafoate; Fluticasone

INTERVENTIONS:
Drug: Tiotropium
Drug: Salmeterol plus Fluticasone

SUMMARY:
The primary objective of this study is to estimate the comparative bronchodilator effect size and variability for tiotropium (Spiriva, 18 µg q.d.) with the free combination of salmeterol (Serevent, 50 µg b.i.d.) and fluticasone (Flixotide, 250 µg b.i.d.) in COPD patients.

International COPD guidelines preserve milder stages of the disease (GOLD stage I and IIa) to bronchodilators and recommend the addition of inhaled corticosteroids only in those patients who have a documented spirometric response to inhaled corticosteroids and in patients with a post-bronchodilator FEV1 of less than 50% predicted, who suffer from frequent exacerbations requiring oral courses of corticosteroids.

Recently published reports indicate that additional bronchodilator efficacy may be achieved when a long-acting beta agonist is combined with an inhaled corticosteroid. Steady state bronchodilation was achieved within one week with the drug combination. However, results of these studies are not consistent, and since the inclusion criteria employed were different from those utilised in the previously conducted tiotropium studies, it is difficult to generalise the observed effects to the general COPD population.

In addition, no comparative data is available on the average response over the 12 daytime hours when COPD patients are active and in most need of bronchodilation. 12 hours corresponds to the dosing intervals for both salmeterol and fluticasone.

DETAILED DESCRIPTION:
This is a six-week, multi-centre, randomised, double-blind, triple-dummy, parallel group pilot study to compare the bronchodilator efficacy and safety of the long-acting bronchodilator tiotropium (Spiriva, 18 µg q.d.) to the free combination of fluticasone (Flixotide, 250 µg b.i.d.) and salmeterol (Serevent, 50 µg b.i.d.) in patients with COPD.

Following an initial screening at Visit 1, subjects will enter a two-week run-in period during which they will record daily rescue salbutamol use in the Patient Daily Diary Card. At Visit 1, pre-dose and post-bronchodilator pulmonary function tests (PFT) will be measured. Four inhalations of ipratropium (20 µg per puff) and four inhalations of salbutamol (100 µg per puff) will be administered 60 minutes prior to obtaining post-bronchodilator PFT measurement.

At Visit 2, a pre-dose PFT will be performed prior to first administration of trial medication. Treatment with blinded study medication (tiotropium or fluticasone + salmeterol) will start in the morning of Visit 2 (Day 1). After three weeks of treatment, at Visit 3 (Day 22), pre-dose FEV1 and FVC will be measured, patient compliance checked and a re-supply of study medication dispensed. After six weeks of treatment, at Visit 4 (Day 43), a 12 hour profile of PFTs will be obtained.

Study Hypothesis:

As this is a pilot trial to investigate the efficacy and safety of tiotropium (18 µg q.d.) as compared to the free combination of fluticasone (250 µg b.i.d.) and salmeterol (50 µg b.i.d.), no formal hypothesis testing will be performed. However, the underlying hypothesis for this trial is that tiotropium is superior to the free combination with respect to the primary efficacy endpoint FEV1AUC0-12 (area under the curve for the time period 0 to 12 hours).

Comparison(s):

At least 100 male or female outpatients with clinical and spirometric evidence of chronic obstructive pulmonary disease (COPD) will be entered in this study. Patients will be randomly assigned to receive either tiotropium inhalation capsules 18 µg q.d., or salmeterol 50 µg oral inhalation b.i.d. in free combination with fluticasone 250 µg oral inhalation b.i.d. in a double-blind triple-dummy fashion.

ELIGIBILITY:
Inclusion criteria:

* All patients must have a diagnosis of chronic obstructive pulmonary disease according to the GOLD criteria and must meet the following spirometric criteria:

  * Patients must have relatively stable airway obstruction with a post-bronchodilator FEV1 < 80% of predicted normal and FEV1/FVC < 70% at Visit 1, and a pre-dose FEV1 < 65% predicted at Visit 2.
* Male or female patients 40 years of age or older. There is no upper age limit.
* Patients must be current or ex-smokers with a smoking history of more than 10 pack-years.

Exclusion criteria:

* Patients with significant diseases other than COPD.
* Patients with a history of asthma, allergic rhinitis or atopy or who have a total blood eosinophil count more than or equal to 600/mm3.
* Patients who have been treated with commercially available tiotropium (Spiriva®).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107
Dates: Start 2003-09; Primary Completion 2004-08 (Actual); Study Completion 2004-08

PRIMARY OUTCOMES:
The primary efficacy endpoint will be FEV1 area under the curve for the time period 0 to 12 hours (FEV1 AUC0-12) measured after 6 weeks of treatment, at the final study visit (Visit 4).

SECONDARY OUTCOMES:
Trough and peak FEV1. Trough FVC at Visits 3 and 4 and peak FVC and FVC AUC0-12 at Visit 4. Individual FEV1 and FVC measurements at each time point. Weekly mean number of puffs of rescue therapy used per day and night.

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. South Africa (Pty.) Ltd.
Locations (12):
- South Africa (12):
  - Tijger Trial Centre, Bellville
  - Boehringer Ingelheim Investigational Site, Bloemfontein
  - UCT Lung Institute, Cape Town
  - Boehringer Ingelheim Investigational Site, Cape Town
  - Durban Lung Centre, Durban
  - St Augustine Hospital, Durban
  - QdotPharma, George
  - Centre for Chest Diseases Research Unit, Johannesburg
  - Boehringer Ingelheim Investigational Site, Paarl
  - Boehringer Ingelheim Investigational Site, Pretoria
  - Vergelegen Medi-Clinic, Somerset West
  - Boehringer Ingelheim Investigational Site, Welkom